CLINICAL TRIAL: NCT02182609
Title: A Phase I Study of Safety, Tolerance, Pharmacokinetics and Nuclear Medicine Imaging of 99mTc-rhAnnexin V-128 Administered Intravenously in Healthy Adult Volunteers
Brief Title: 99mTc-rhAnnexin V-128: a First In Man Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Collaborators: Atreus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001; CAAA113A12101 (Other: Novartis)
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 99mTc-rhAnnexin V-128 (Experimental)
  Interventions: Drug: Kit for the Preparation of 99mTc-rhAnnexin V-128

INTERVENTIONS:
Drug: Kit for the Preparation of 99mTc-rhAnnexin V-128 — Kit for the Preparation of Tc-99m Recombinant Human Annexin V-128 for Injection

SUMMARY:
The objectives of this study are:

* To determine the safety and tolerability of a single dose of 99mTc-rhAnnexin V-128 administered as an intravenous bolus over 10-20 seconds.
* To determine the biodistribution, pharmacokinetics and radiation dosimetry of 99mTc-rhAnnexin V-128 in normal healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. No significant medical history
3. Normal physical examination
4. No clinically significant abnormalities in baseline laboratory values
5. No clinically significant abnormalities on 12 lead electrocardiogram
6. Female subjects must be post-menopausal, surgically sterilized or have negative urine beta human chorionic gonadotropin pregnancy test at initial screening and pre-injection on dosing day
7. Written informed consent signed

Exclusion Criteria:

1. Pregnancy or lactation
2. Know hypersensitivity to the investigational drug or any of its components
3. Current enrolment in another investigational study
4. Unwillingness to provide or continue informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | Whole study period
  Type and incidence of AEs, as well as severity and relatedness to the study medication will be tabulated. Special attention will be given to those subjects who prematurely discontinue the study or the study medication due to an AE, or who experience a severe AE or an SAE.
Laboratory assessments | baseline and 24 hrs, 72 hrs and 30 days after injection
  Laboratory data (Hematology, coagulation, biochemistry, and urinalysis) will be analysed with respect to the normal ranges of values provided by the local laboratory and with respect to pre-defined levels of change in these values.
  Abnormal laboratory test results will be tabulated.
Electrocardiography | screening and immediatly, 24hrs, 72 hrs, 7 days and 30 days after injection
  ECG parameters will include heart rate (HR), RR interval, PR interval, QRS width and QT interval.
  ECG results will be evaluated by means of descriptive statistics and frequency tabulations.
Vital signs | At each study visit
  Descriptive statistics of the vital signs (pulse rate and blood pressure) observed values as well as for the changes from baseline value will be created. Frequency tabulations with values within, below or above the normal ranges will be made.

SECONDARY OUTCOMES:
rhAnnexin V-128 serum concentration | 0, 5, 10, 15, 30, 60, 90, minutes and 3 h, 6h and 24 h post-injection
  In addition to dosimetry, pharmacokinetic will be assessed based on rhAnnexin V-128 serum concentration
Whole-body SPECT imaging | 30min, 90min, 3hrs, 6hrs and 24 hours post-injection
  The quantitative in vivo biodistribution (whole body dosimetry) of the 99mTc-rhAnnexin V-128 will be determined through whole-body SPECT imaging.
Blood sample counting | baseline and 0, 5,10, 15, 30, 60, 90 min, 3 h, 6 h and 24 hours post-injection
  Radioactivity of the whole blood and serum samples will be counted in a gamma counter to assess blood dosimetry and pharmacokinetic.
Amount of 99mTc excreted in urine | One sample at baseline and urine collection within 24 hours post-injection
Amount of 99mTc excreted in faeces | Baseline and within 24h post injection
Anti-rhAnnexin V-128 IgG and IgM antibodies | Baseline and 14 and 30 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D. Rudy, MD, FRCPC, Principal Investigator — The University of Ottawa Heart Institute, The Ottawa Hospital
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada